CLINICAL TRIAL: NCT04305522
Title: A Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Two Probiotic Interventions For The Prophylaxis of Migraine in Patients Diagnosed With Episodic Migraine
Brief Title: Probiotics for the Prophylaxis of Migraine
Acronym: MIGR_PRO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIGR_PRO.2
Record Dates: First submitted 2020-03-03; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Migraine
Keywords: Probiotic; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic 1 group (Experimental): A commercially-available multi-strain probiotic with added magnesium and vitamin B6
  Interventions: Dietary Supplement: Probiotic 1
- Probiotic 2 group (Experimental): A multi-strain probiotic
  Interventions: Dietary Supplement: Probiotic 2
- Placebo group (Placebo Comparator): Identical placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic 1 — Probiotic mixture with maltodextrin as a carrier.
  Arms: Probiotic 1 group
Dietary Supplement: Placebo — Placebo comparator with maltodextrin as a carrier.
  Arms: Placebo group
Dietary Supplement: Probiotic 2 — Probiotic mixture with maltodextrin as a carrier.
  Arms: Probiotic 2 group

SUMMARY:
This study aims to understand the efficacy of two probiotic interventions as prophylaxes of migraine symptoms in individuals diagnosed with episodic migraine.

The primary outcome measure will be migraine days per month, but secondary outcome measures such as use of analgesia, the wider impact of migraine (as assessed through the HIT-6 score) will also be assessed. Finally adverse effects will be evaluated.

The study will have three arms: two arms including the two different probiotic preparations and a third placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 65 years.
2. Signature of informed consent by the patient.
3. Patients with confirmed migraine, diagnosed by a neurologist
4. Patient-indicated frequency of migraine attacks (or days) of at least 4 per month.
5. Fairly predictable and stable pattern of migraine attacks (frequency, duration, intensity)

Exclusion Criteria:

1. Patients diagnosed with chronic migraine
2. Migraine patients suffering from medication-dependent headaches.
3. Patients suffering from cluster or tension-related headaches.
4. Patients who used antibiotics up to two weeks before the start of the study.
5. Patients who have taken other probiotics in the previous two months.
6. Patients with chronic use of non-steroidal anti-inflammatory drugs.
7. Patients with inflammatory bowel disease (due to increased intestinal permeability).
8. Patients who are pregnant, breastfeeding or who do not commit to using an effective method of contraception during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-02-02 (Estimated); Study Completion 2021-05-02 (Estimated)

PRIMARY OUTCOMES:
Number of days with migraine episodes | 4-week
  Number of days with migraine episodes in weeks 4
Number of days with migraine episodes | 8-week
  Number of days with migraine episodes, in weeks 8
Number of days with migraine episodes | 12-week
  Number of days with migraine episodes, in weeks 12.

SECONDARY OUTCOMES:
Number of migraine episodes | 4 weeks
  Number of migraine episodes, in weeks 4
Number of migraine episodes | 8 weeks
  Number of migraine episodes, in weeks 8
Number of migraine episodes | 12 weeks
  Number of migraine episodes, in weeks 12.
Number of days that each patient requires the administration analgesia | 4 weeks
  Number of days that each patient requires the administration analgesia, in weeks 4
Number of days that each patient requires the administration analgesia | 8 weeks
  Number of days that each patient requires the administration analgesia, in weeks 8
Number of days that each patient requires the administration analgesia | 12 weeks
  Number of days that each patient requires the administration analgesia, in weeks 12
Headache Impact Test (HIT-6) score | 4 weeks
  Headache Impact Test (HIT-6) score at weeks 0 and 4 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Headache Impact Test (HIT-6) score | 8 weeks
  Headache Impact Test (HIT-6) score at weeks 8 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Headache Impact Test (HIT-6) score | 12 weeks
  Headache Impact Test (HIT-6) score at weeks 12 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Treatment adherence rate | 12 weeks
  Treatment adherence rate using the returned capsules.
Number of adverse events | 12 weeks
  Numbre od adverse effects reported
Adherence to the treatment. | 12 weeks
  Percentage of treatment intake days.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante

IPD SHARING:
Plan to Share IPD: No